CLINICAL TRIAL: NCT06528977
Title: Effects of a 10-day Western Diet on Cardiometabolic and Immune Function in Midlife Adults
Brief Title: Western Diet on Cardiometabolic and Immune Function
Acronym: WD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2199946; P20GM113125 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Aging; Diet, Healthy
Keywords: added sugars; western diet; cardiometabolic health; T-cell function; intestinal permeability
MeSH Terms: interventions — Diet, Western

STUDY DESIGN:
Intervention Model Description: A controlled feeding study prepared by registered dieticians. Participants will be pre-tested, provided a 10-day WD to be tested on day 10, then post-tested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Western Diet (Experimental): Consumption of 10 days of a diet high in added sugars (25% of total caloric intake)
  Interventions: Other: Western Diet

INTERVENTIONS:
Other: Western Diet — Consumption of 10 days of a diet high in added sugars (25% of total caloric intake)

SUMMARY:
This study will implement a Western Diet (WD) to understand cardiometabolic and immune function in middle-aged adults (50- 64 years old). Vascular health, intestinal permeability, and T-cell function will be examined before, during, and after the WD. The WD is a 10-day diet and will consist of 25% of total energy from added sugars.

DETAILED DESCRIPTION:
Aging is the primary risk factor for Alzheimer's disease (AD) which is the most common form of dementia and among the fastest-growing causes of morbidity and mortality in the United States. The risk factors for AD emerge during midlife and are similar to cardiovascular diseases, one of which has particular interest is high blood pressure. The impact of blood vessels and high blood pressure are made worse by poor lifestyle habits, including eating a Western Diet (WD) that contains processed food and high amounts of added sugars (e.g., foods containing high amounts of fructose), with little to no fiber intake from fruits and vegetables. Previous data indicates a 10-day WD can acutely increase triglycerides and blood pressure. These cardiometabolic changes are thought to involve the immune system, however, it is not exactly known how a WD triggers an inflammatory response. This project aims to determine the role of diet-induced changes in gut health and the function of the immune system (T-cells) in midlife adults. It is hypothesized that eating a WD will acutely make the small intestine more permeable, concurrent with activation of the immune system measured via T-cell function. To test this hypothesis, gut health, T-cell function, and blood vessel function will be measured before, during, and after a 10-day WD. The data generated from this project will help bridge the gap in understanding the relation between diet and the immune system. The results will support future grant proposals to the National Institutes of Health aimed at using dietary interventions to protect against high blood pressure and cognitive impairment in mid-life adults.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent
* men and postmenopausal women aged 50-64 years
* systolic blood pressure < 130 mmHg; diastolic blood pressure < 90 mmHg
* body mass index (BMI) <30 kg/m2 and % body fat < 25% for men and < 33% for women
* fasting triglycerides < 200 mg/dl (< 2.3 mmol/L)
* low density lipoprotein (LDL) cholesterol <160 mg/dl (4.14 mmol/L)
* fasting plasma glucose <126 mg/dl (<7.0 mmol/L)
* weight stable in the prior 6 months (≤ 2 kg weight change)
* blood chemistries indicative of normal liver enzymes and renal function (estimated glomerular filtration rate using the Modification of Diet in Renal Disease (MDRD) prediction equation must be >60 ml/min/1.73 m^2)

Exclusion Criteria:

* current use of medications or supplements known to lower blood triglycerides or cholesterol (e.g., fibrates, statins, high dose niacin, high dose omega-3 supplement)
* chronic clinical diseases (e.g., coronary artery/peripheral artery/cerebrovascular diseases, heart failure, diabetes, chronic kidney disease requiring dialysis, neurological or autoimmune conditions affecting cognition (e.g. Alzheimer's disease or other forms of dementia, Parkinson's disease, epilepsy, multiple sclerosis, large vessel infarct)
* major psychiatric disorder (e.g. schizophrenia, bipolar disorder)
* current or past (i.e., last 3 months) use of anti-hypertensive or other cardiovascular-acting medications known to influence vascular function and/or arterial stiffness
* current medication use likely to affect central nervous system (CNS) functions (e.g. long active benzodiazepines)
* concussion within last 2 years and ≥ 3 lifetime concussions
* heavy alcohol consumption (≥8 drinks/week for women and ≥15 drinks/week for men)
* recent major change in health status within the previous 6 months (i.e., surgery, significant infection, or illness)
* current smoking within the past 3 months.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Arterial Blood Pressure (mmHg) | Over the course of 1-2 months
  Comparison between before, during and after western diet
Change in relative brachial artery flow-mediated dilation (%) | Over the course of 1-2 months
  Comparison between before, during and after western diet
Change in absolute brachial artery flow-mediated dilation (mm) | Over the course of 1-2 months
  Comparison between before, during and after western diet
Change in T-cell mitochondria respiration (oxygen consumption rate) | Over the course of 1-2 months
  Comparison between before, during and after western diet
Change in T-cell flow cytometry (%) | Over the course of 1-2 months
  Comparison between before, during and after western diet
Change in intestinal permeability (lactulose : mannitol test) | Over the course of 1-2 months
  Comparison between before, during and after western diet
Change in triglycerides (mg/dL) | Over the course of 1-2 months
  Comparison between before, during and after western diet
Change in cholesterol (mg/dL) | Over the course of 1-2 months
  Comparison between before, during and after western diet

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Martens, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No